CLINICAL TRIAL: NCT05950308
Title: Assessment of Immune Response in Multiple Sclerosis Patients With COVID-19/Vaccination Treated With Ofatumumab and Other Disease Modifying Therapies
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GUS23
Record Dates: First submitted 2023-07-14; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- HC: Healthy control
- OFA: Received ofatumumab
- OCR: Received ocrelizumab
- S1P: Received sphingosine-1-phosphate receptor modulator

SUMMARY:
Vaccine responses in patients treated with anti-CD20 antibodies (ocrelizumab and ofatumumab) or S1P receptor modulators (fingolimod and siponimod) were evaluated before and after third SARS-CoV-2 vaccination as part of an ongoing longitudinal study. Total spike protein and spike receptor binding domain (RBD)-specific immunoglobulin G (IgG) responses were measured by Luminex bead-based assay. Spike-specific CD4+ and CD8+ T cell responses were measured by activation-induced marker expression.

ELIGIBILITY:
Inclusion Criteria

All Participants:

* Aged 18-75 years old MS Patients
* Diagnosed with MS based on 2017 McDonald criteria

Exclusion Criteria

All Participants:

* Participants with a known history of COVID-19 Healthy Adults
* Immunocompromised or on immunosuppressive therapy MS Patients
* None specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving humoral response (i.e. immune response) to an FDA-authorized COVID 19 vaccine in ofatumumab treated participants | varied up to 6 months
Percentage of participants achieving T-cell response (i.e. immune response) to an FDA-authorized COVID 19 vaccine in ofatumumab treated participants | varied up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States